CLINICAL TRIAL: NCT03245671
Title: Particulate vs. Nonparticulate Epidural Steroid Injections for the Treatment of Symptomatic Unilateral Lumbar Foraminal Stenosis: a Prospective Double-blinded Randomized Study
Brief Title: Particulate vs. Nonparticulate Epidural Steroid Injections for Lumbar Foraminal Stenosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to address regulatory concerns.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0615
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — dexamethasone 21-phosphate; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Decadron (Active Comparator): Patients in the Decadron group will receive epidural injections containing a total of 15 mg Decadron.
  Interventions: Drug: Decadron Phosphate, Injectable; Procedure: Epidural Steroid Injection
- Kenalog (Active Comparator): Patients in the Kenalog group will receive epidural injections containing a total of 80 mg Kenalog.
  Interventions: Drug: Kenalog Injectable Product; Procedure: Epidural Steroid Injection

INTERVENTIONS:
Drug: Kenalog Injectable Product — 80 mg of Kenalog will be used.
  Arms: Kenalog
Drug: Decadron Phosphate, Injectable — 15 mg of Decadron will be used.
  Arms: Decadron
Procedure: Epidural Steroid Injection — Patient will receive epidural steroid injections of either Kenalog or Decadron.

SUMMARY:
Chronic lumbosacral radiculopathy secondary to lumbar spinal stenosis affects a large number of individuals, and there is a general lack of consensus in the medical community in terms of effective treatments for this problem. By assessing the relative efficacy of transforaminal epidural injections of particulate and nonparticulate steroids, this study attempts to further define the appropriate conservative management of painful unilateral radiculopathies due to unilateral lumbar foraminal stenosis. Patients will be randomized to receive a transforaminal epidural injection of either a particulate (Kenalog) or nonparticulate (Decadron) steroid. Outcomes will be assessed at 2 weeks, 6 weeks, 3 months, and 6 months following the injection.

ELIGIBILITY:
Inclusion Criteria:

* English speaking/reading adults age 18-90 years
* Patients with complaints of unilateral radicular lower extremity symptoms
* NRS pain score >= 5
* Pain symptoms for at least 1 month's duration
* Patients deemed appropriate for lumbar transforaminal epidural steroid injections by treating spine specialist
* Targeted injection level for L4 or L5
* MRI of lumbosacral spine that demonstrates and confirms single-level neural compression secondary to unilateral lumbosacral foraminal or subarticular stenosis consistent with clinical history and findings
* Lumbar foraminal stenosis severity of grades 1, 2, and 3

Exclusion Criteria:

* Patients with multiple symptomatic levels
* Patients who are deemed not appropriate to undergo lumbar transforaminal epidural steroid injections (e.g., allergy to local anesthetics, radiographic dye contrast, patients with high bleeding tendency, pregnancy)
* Patients involved with litigation or worker's compensation cases
* Patients who are unable to answer the questionnaires and perform follow-up visits
* Patients who have active, concurrent painful diagnoses (e.g., hip osteoarthritis, greater trochanteric pain syndrome, knee pain, peripheral vascular disease, or peripheral neuropathy) that may confuse clinical picture and impact patients' rating and perception of their low back and radicular symptoms
* Patients with other spinal pathologies confirmed on imaging that may explain patient's pain
* Patients who have additional severe foraminal stenosis inferior to the symptomatic level (e.g., symptomatic L4 foraminal stenosis with severe L5 foraminal stenosis) will not have those levels injected
* Non-English speakers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Improvement in function (2 weeks post-injection) | 2 weeks post-injection
  This will be measured using the Oswestry Disability Index (ODI; 0-100 scale). A higher score represents greater disability (greater pain and functional limitations).
Improvement in function (6 weeks post-injection) | 6 weeks post-injection
  This will be measured using the ODI (0-100 scale). A higher score represents greater disability (greater pain and functional limitations).
Improvement in function (3 months post-injection) | 3 months post-injection
  This will be measured using the ODI (0-100 scale). A higher score represents greater disability (greater pain and functional limitations).
Improvement in function (6 months post-injection) | 6 months post-injection
  This will be measured using the ODI (0-100 scale). A higher score represents greater disability (greater pain and functional limitations).

SECONDARY OUTCOMES:
Medication use | 2 weeks, 6 weeks, 3 months, and 6 months post-injection
  The use of any pain medications (e.g., opioids, anti-inflammatory drugs, neuropathic medications) will be collected.
Patient satisfaction with the procedure | 2 weeks, 6 weeks, 3 months, and 6 months post-injection
  Satisfaction will be assessed using the North American Spine Society Outcome Questionnaire. Patients will be asked to pick from 4 multiple choice statements regarding their satisfaction with their procedure.
Quality of life | 2 weeks, 6 weeks, 3 months, and 6 months post-injection
  This will be assessed using the Veterans RAND 12-item Health Survey.
Side effects | 2 weeks, 6 weeks, 3 months, and 6 months post-injection
  Side effects, including bleeding, infection, allergic reaction, dural puncture, nerve damage, and paralysis, will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States